CLINICAL TRIAL: NCT07122271
Title: Joint Effects of Physical Activity and Diet Quality on Depression and Mortality in U.S. Adults With Diabetes: A Population-Based Cohort Study Using NHANES 2007-2018 With Mediation and Machine Learning Analyses
Brief Title: Joint Effects of Physical Activity and Diet Quality on Depression and Mortality in Diabetes
Status: Completed | Type: Observational
Sponsor: Minghui Wang (Other)
Responsible Party: Sponsor-Investigator, Minghui Wang, Principal Investigator, Wuhan Sports University
Organization: Wuhan Sports University (Other)
Other Study IDs: WuhanSU
Record Dates: First submitted 2025-08-03; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Complications; Depression Anxiety Disorder; Diabetes
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 120 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to investigate whether physical activity (PA) and diet quality (DQ) can reduce depression and mortality risk in individuals with diabetes. Participants will be adults diagnosed with diabetes during the 2007-2018 cycle of the National Health and Nutrition Examination Survey (NHANES). The main questions to be answered include:

Does higher levels of physical activity significantly reduce the risk of depression in individuals with diabetes? Is higher diet quality associated with lower mortality in individuals with diabetes? Investigators will compare individuals with varying levels of PA and DQ to examine whether these two lifestyle factors, both individually and in combination, have protective effects on mental health and survival.

Participants will:

Complete questionnaires regarding their physical activity and dietary intake; Be assessed for depressive symptoms (PHQ-9); Be enrolled in long-term mortality follow-up (from the National Death Index); Analyses will be categorized according to their PA (measured in MET-min/week) and HEI-2015 dietary score.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 years and older.
* Diagnosed with diabetes mellitus, defined by self-report, fasting plasma glucose ≥126 mg/dL, or HbA1c ≥6.5%.
* Available data on physical activity, diet quality (HEI-2015), and depression status (PHQ-9).
* Complete demographic and mortality follow-up data.

Exclusion Criteria:

* Missing key exposure or outcome data (e.g., physical activity, HEI-2015, PHQ-9, mortality).
* Pregnant individuals at the time of the survey.
* Participants with unreliable or extreme dietary intake data (e.g., energy intake <500 or >5000 kcal/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult participants aged 20 years and older with a confirmed diagnosis of diabetes mellitus from the NHANES 2007-2018 dataset. The population comprises individuals with available data on physical activity, diet quality, and depression symptoms, as well as complete demographic and mortality information. Participants represent a nationally representative sample of the non-institutionalized US population.
  Subgroup analyses were conducted by sex, age group, and BMI category to explore potential effect modification.Machine learning and mediation analysis were also applied to further explore the underlying mechanisms and effect modification.
Sampling Method: Probability Sample
Enrollment: 3621 (Actual)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Proportion of Adults With Diabetes Meeting Depression Criteria at Baseline (PHQ-9 ≥5) | At the time of baseline NHANES examination for each 2-year survey cycle, including 2007-2008, 2009-2010, 2011-2012, 2013-2014, 2015-2016, and 2017-2018 (6 cycles in total, each lasting 2 years).
  Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item self-report instrument scored from 0 to 27. Participants scoring ≥5 will be classified as having depressive symptoms. The outcome is the percentage of participants who meet this criterion at baseline.

SECONDARY OUTCOMES:
Odds Ratio for Depression by Physical Activity Category in Adults With Diabetes | At the time of baseline NHANES examination for each 2-year survey cycle, including 2007-2008, 2009-2010, 2011-2012, 2013-2014, 2015-2016, and 2017-2018 (6 cycles in total, each lasting 2 years).
  Physical activity will be assessed using NHANES physical activity questionnaires and expressed in metabolic equivalent minutes per week (MET-min/week). Participants will be categorized into three PA levels: inactive (<600 MET-min/week), insufficiently active (600-1,199 MET-min/week), and sufficiently active (≥1,200 MET-min/week). Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item self-report instrument scored from 0 to 27, with scores ≥5 indicating the presence of depressive symptoms. Logistic regression models will be used to estimate odds ratios for depression across PA categories, using the inactive group as the reference.Odds Ratio (95% Confidence Interval)
Odds Ratio for Depression by Diet Quality Category in Adults With Diabetes | At the time of baseline NHANES examination for each 2-year survey cycle, including 2007-2008, 2009-2010, 2011-2012, 2013-2014, 2015-2016, and 2017-2018 (6 cycles in total, each lasting 2 years).
  Diet quality will be assessed using the Healthy Eating Index-2015 (HEI-2015) score, derived from two 24-hour dietary recall interviews. Scores range from 0 to 100, with higher scores indicating better diet quality. Participants will be categorized into two groups: unqualified diet quality (HEI-2015 <60) and qualified diet quality (HEI-2015 ≥60). Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item self-report instrument scored from 0 to 27, with scores ≥5 indicating the presence of depressive symptoms. Logistic regression models will be used to estimate odds ratios for depression between diet quality groups, using the unqualified group as the reference.Odds Ratio (95% Confidence Interval)
Odds Ratio for Depression by Combined Physical Activity and Diet Quality Categories in Adults With Diabetes | At the time of baseline NHANES examination for each 2-year survey cycle, including 2007-2008, 2009-2010, 2011-2012, 2013-2014, 2015-2016, and 2017-2018 (6 cycles in total, each lasting 2 years).
  Physical activity (PA) will be assessed using NHANES physical activity questionnaires and expressed in metabolic equivalent minutes per week (MET-min/week). Diet quality (DQ) will be assessed using the Healthy Eating Index-2015 (HEI-2015) score, derived from two 24-hour dietary recall interviews. Participants will be classified into four PA_DQ groups:
  Inactive_Unqualified (PA <600 MET-min/week and HEI-2015 <60) Inactive_Qualified (PA <600 MET-min/week and HEI-2015 ≥60) Active_Unqualified (PA ≥600 MET-min/week and HEI-2015 <60) Active_Qualified (PA ≥600 MET-min/week and HEI-2015 ≥60) Depression will be measured using the Patient Health Questionnaire-9 (PHQ-9), a validated 9-item self-report instrument scored from 0 to 27, with scores ≥5 indicating the presence of depressive symptoms. Logistic regression models will be used to estimate odds ratios for depression across the four PA_DQ groups, using the Inactive_Unqualified group as the reference.Odds Ratio (95% Confidence Interval)
Subgroup analysis for All-Cause Mortality by Combined Physical Activity and Diet Quality Categories in Adults With Diabetes and Comorbid Depression | From baseline NHANES examination to December 31, 2019 (up to 120 months follow-up)
  All-cause mortality will be determined from the NHANES Linked Mortality Files, which are linked to the National Death Index (NDI). Participants will be classified into four combined PA_DQ categories:
  Inactive_Unqualified (PA <600 MET-min/week and HEI-2015 <60) Inactive_Qualified (PA <600 MET-min/week and HEI-2015 ≥60) Active_Unqualified (PA ≥600 MET-min/week and HEI-2015 <60) Active_Qualified (PA ≥600 MET-min/week and HEI-2015 ≥60) Subgroup analyses will examine whether hazard ratios for all-cause mortality associated with these PA_DQ categories differ across age (<65 vs ≥65 years), sex, BMI (<29 vs ≥29 kg/m²), and sedentary time (<4 vs ≥4 hours/day). Cox proportional hazards models with interaction terms will be used, and results will be reported as stratified hazard ratios relative to the Inactive_Unqualified group.

OTHER OUTCOMES:
SHAP Analysis of Key Predictors of Depression Risk in Adults With Diabetes | At the time of baseline NHANES examination for each 2-year survey cycle, including 2007-2008, 2009-2010, 2011-2012, 2013-2014, 2015-2016, and 2017-2018 (6 cycles in total, each lasting 2 years).
  Shapley Additive exPlanations (SHAP) analysis will be used to identify and rank the most important predictors of depression risk, defined as Patient Health Questionnaire-9 (PHQ-9) score ≥5. Predictors assessed will include physical activity (PA), diet quality (DQ), body mass index (BMI), education, poverty-income ratio (PIR), age, sex, and sedentary behavior. Results will be reported as variable importance rankings with SHAP values.Relative importance score (SHAP value).
Mediation Effect of BMI on the Association Between Combined Physical Activity and Diet Quality and Depression in Adults With Diabetes | At the time of baseline NHANES examination for each 2-year survey cycle, including 2007-2008, 2009-2010, 2011-2012, 2013-2014, 2015-2016, and 2017-2018 (6 cycles in total, each lasting 2 years).
  Causal mediation analysis will be used to estimate the indirect effect of body mass index (BMI, kg/m²) on the association between combined physical activity and diet quality (PA_DQ) and depression, defined as Patient Health Questionnaire-9 (PHQ-9) score ≥5. Participants will be classified into four PA_DQ categories:Inactive_Unqualified (PA <600 MET-min/week and HEI-2015 <60),Inactive_Qualified (PA <600 MET-min/week and HEI-2015 ≥60),Active_Unqualified (PA ≥600 MET-min/week and HEI-2015 <60)
  ,Active_Qualified (PA ≥600 MET-min/week and HEI-2015 ≥60).The outcome will be reported as the average causal mediation effect (ACME) and the proportion mediated (%), using the Inactive_Unqualified group as the reference category.Average Causal Mediation Effect (ACME) and proportion mediated (%)

CONTACTS AND LOCATIONS:
Overall Officials: zeng chen, Principal Investigator — Geriatric Hospital of Hainan province
Locations (1):
- Wuhan Sports University, Wuhan, Hubei, China

REFERENCES:
- See also: Related Info — https://wwwn.cdc.gov/Nchs/Data/Nhanes/Public/2007/DataFiles/PAQ_E.htm
- See also: Related Info — https://www.cdc.gov/nchs/nhanes/